CLINICAL TRIAL: NCT06639815
Title: Evaluation of Tooth Development in Molar Incisor Hypomineralization with Cameriere and Haavikko Methods for Dental Age Estimation: a Case-control Study
Brief Title: Tooth Development in Molar Incisor Hypomineralisation
Status: Completed | Type: Observational
Sponsor: Canan Bayraktar Nahir (Other)
Responsible Party: Sponsor-Investigator, Canan Bayraktar Nahir, Assistant Professor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Other Study IDs: 23-KAEK-113
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Molar Incisor Hypomineralization
Keywords: children; dental age estimation; dental development
MeSH Terms: conditions — Molar Hypomineralization | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: with molar incisor hypomineralization
  Interventions: Other: clinical and radiographic examination
- Group 2: without molar incisor hypomineralization
  Interventions: Other: clinical and radiographic examination

INTERVENTIONS:
Other: clinical and radiographic examination — clinical and radiographic examination

SUMMARY:
Molar incisor hypomineralization has been defined as a qualitative developmental enamel defect affecting one or more permanent first molars, often including the permanent incisors. The development of the teeth with the developmental defect remains unclear.

The aim of this study is to evaluate tooth development in children with MIH using the Cameriere and Haavikko methods on panoramic radiographs and to determine the accuracy of these methods. The first null hypothesis of this study was that there would be no difference in tooth development between children with MIH and children with healthy structure of teeth, and the second null hypothesis was that Cameriere and Haavikko methods could estimate dental age with the equal accuracy.

DETAILED DESCRIPTION:
This study was planned to evaluate tooth development in a cohort of 8- to 12-year-old children diagnosed with MIH who applied to the Department of Pedodontics, Faculty of Dentistry, Tokat Gaziosmanpaşa University, for dental examinations or treatment between June 1, 2023, and June 1, 2024.

The study group (Group 1) was determined according to gender and chronological age group from children who were diagnosed with MIH as a result of dental examination and met the inclusion criteria. The control group (Group 2) was selected from children matched to MIH cases according to gender and chronological age, without signs of hypomineralisation and met the inclusion criteria.

The chronological age of the children was calculated using Microsoft Excel 2013 (Microsoft, Redmond, WA, USA). The following formula was applied:

"[(date of panoramic radiography) - (documented date of birth)] / 365.25" Tooth development was determined on panoramic radiographs taken with a single device (J. Morita Mfg. Corp., Kyoto, Japan) using the Cameriere and Haavikko methods.

The data were analyzed using the IBM Statistical Package for the Social Sciences (SPSS for Windows, version 26.0, SPSS Inc., Chicago, IL, USA). Data from the two dental age estimation methods were analyzed for each gender and age group within Group 1 and Group 2. The Kolmogorov-Smirnov test was applied to assess normality. The Spearman correlation coefficient was employed to examine the relationship between chronological and dental age, and the Paired Samples T-test and Wilcoxon Signed-rank Test were used to compare the difference. The Independent Samples T-test and Mann-Whitney U test were utilized to compare chronological and dental age based on MIH presence. Intraclass Correlation Coefficient (ICC) was calculated to assess inter- and intra-observer reliability. Quantitative data are presented as mean ± standard deviation and median (minimum-maximum), while categorical data are presented as frequency (percentage). Statistical significance was set at the 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

must have parental consent must have high-quality panoramic radiographs

Exclusion Criteria:

systemic disease tooth agenesis hyperdontia

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who apply to Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Pedodontics due to any dental problem.
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Tooth development | 1 day
  Distribution of children according to the group, chronological age and gender Evaluation of dental development of Group 1 and 2 according to gender and dental age estimation methods Comparison of chronological age and dental age estimated by two different dental age estimation methods according to groups and gender Comparison of chronological age and dental age according to different dental age methods, chronological age groups and presence of MIH in girls Comparison of chronological age and dental age according to different dental age methods, chronological age groups and presence of MIH in boys The agreement between dental age and chronological age in Group 1 and 2 according to gender and dental age estimation methods

CONTACTS AND LOCATIONS:
Overall Officials: Esra Ergün, Research Assistant, Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Tokat Gaziosmanapaş University, Tokat Province, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
with the link to be prepared later

REFERENCES:
- [Background] Tunc ES, Ulusoy AT, Bayrak S, Cankaya S. Dental development in children with severe molar-incisor hypomineralization in Samsun, Turkey. J Oral Sci. 2013 Sep;55(3):203-7. doi: 10.2334/josnusd.55.203. PMID 24042586
- See also: Tunc ES, Ulusoy AT, Bayrak S, Cankaya S. Dental development in children with severe molar-incisor hypomineralization in Samsun, Turkey. J Oral Sci 2013;55:203-207. — https://pubmed.ncbi.nlm.nih.gov/24042586/